CLINICAL TRIAL: NCT06792487
Title: Analysis of the Immune Infiltrate in Lesional Skin During Anti-interleukin 23 (IL-23) Therapy in Patients With Moderate-severe Plaque Psoriasis
Brief Title: Immune Infiltrate Analysis of Psoriasis Skin During Therapy With Anti-interleukin 23 (IL-23)
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6215
Record Dates: First submitted 2024-01-26; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sperimental: Patients affected by moderate-severe psoriasis treated with anti IL-23 therapy for at least 6 months, according to label dose.
  Interventions: Procedure: skin biopsy
- No Sperimental: Patients affected by moderate-severe psoriasis that have not been already treated
  Interventions: Procedure: skin biopsy

INTERVENTIONS:
Procedure: skin biopsy — punch biopsy (6 mm) of lesional psoriasis skin

SUMMARY:
Psoriasis is an immune-mediated inflammatory skin disease characterized by the presence of erythematous and itchy plaques.

Psoriasis has a multifactorial pathogenesis, environmental and genetic factors contribute to its development.

Although interleukin-23 blockade has been shown to be highly effective in the treatment of psoriasis, relapses have occurred during therapy.

Our study aims to identify the cellular source of key cytokines involved in disease recurrence or persistence of at least one psoriatic lesion in patients affected by moderate- severe psoriasis treated with an anti-IL-23 biologic drug. The immune infiltrate of resistant or relapsed plaques during anti-IL-23 therapy will be analysed from skin biopsies.

ELIGIBILITY:
Inclusion Criteria:

* moderate-severe psoriasis PASI>10
* anti IL 23 biologic therapy for at least 6 months (for the group under treatment)
* during therapy at least one area resistant to treatment or at least one flare of disease (for the group under treatment)
* patients able to express informed consent

Exclusion Criteria:

* patients unable to express informed consent
* patients with complete response to anti IL23, without resistant plaques or disease flare-ups

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients affected by moderate-severe psoriasis under anti IL-23 therapy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Identify the cellular source of key cytokines involved in disease recurrence or persistence of at least a psoriatic lesion | through study completion, an average of 1 year
  Through the integration of multiparametric immunofluorescence staining with RNA in situ hybridization technology, our study aims to identify the cellular source of key cytokines involved in disease recurrence or persistence of at least one lesion psoriatic lesion in patients with moderate-severe psoriasis, undergoing treatment with anti-IL-23.

SECONDARY OUTCOMES:
immune biomarkers of sustained and prolonged response to treatment | through study completion, an average of 1 year
  Identification of possible immune biomarkers of sustained and prolonged response to anti-IL-23 biological therapy that will include the expression profile of biomarkers related to tissue immune memory.

CONTACTS AND LOCATIONS:
Overall Officials: Ketty Peris, Prof, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC Dermatologia, Rome, Lazio, Italy